CLINICAL TRIAL: NCT02849574
Title: Evaluation of Changes in Consumption of Drugs and Substances After Incarceration
Acronym: COSMOS
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC14_0259
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Addictions
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To improve the management and risk reduction, it is essential to understand the evolution of the consumption of psychoactive substances, medicated or not in detention; it does not have at present no data on this subject. This work has as main objective to evaluate the development of substance use terms (goods and consumption practices) by the inmates between the period preceding their incarceration and their fifth month in detention.

ELIGIBILITY:
Inclusion Criteria:

* Major subject
* Subject in the fourth or fifth month of incarceration
* Held about agreeing to participate in the study

Exclusion Criteria:

* Patient refusing to participate
* Patient unable to respond to the questionnaire (major difficulties understanding of the French language)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligible study population is incarcerated major subjects. The topics will be selected subjects incarcerated in remand centers participating in the study. All subjects were medical examination, Home Maintenance arriving at their entrance into custody. On this occasion, the medical staff will verify the absence of non inclusion criterion and the subject will be informed orally and via an information sheet that will retain an invitation to respond to an anonymous questionnaire will be sent after him 4 or 5 months of detention (as prisons). He may accept or reject this invitation.
Sampling Method: Non-Probability Sample
Enrollment: 629 (Actual)
Dates: Start 2015-01; Primary Completion 2015-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
change in practices of consumption of psychoactive substances between the period prior to incarceration and detention period | Until 5 months
  composite endpoint representing the existence of a change in practices of consumption of psychoactive substances between the period prior to incarceration and detention period

CONTACTS AND LOCATIONS:
Overall Officials: Caroline VICTORRI-VIGNEAU, Dr, Principal Investigator — Nantes University Hospital
Locations (6):
- France (6):
  - Angers University Hospital, Angers
  - Fontenay Le Comte Hospital, Fontenay-le-Comte
  - La Roche sur Yon Hospital, La Roche-sur-Yon
  - Laval Hospital, Laval
  - Le Mans Hospital, Le Mans
  - Nantes University Hospital, Nantes

IPD SHARING:
Plan to Share IPD: No